CLINICAL TRIAL: NCT02461121
Title: Compare the Safety and Effective of HLA-mismatched Microtransplantation With HLA-matched Nonmyeloablative Transplantation for Acute Myeloid Leukemia in Intermediate-risk
Brief Title: HLA-mismatched MST vs HLA-matched NST for AML in Intermediate-risk
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MST vs NST
Record Dates: First submitted 2015-05-18; First posted 2015-06-03 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; microtransplantationHLA-mismatched microtransplantation; nonmyeloablative stem cell transplantation; graft-versus-host disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Graft vs Host Disease | interventions — Cyclosporine; Mycophenolic Acid; Cytarabine; fludarabine; Antilymphocyte Serum; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MST（microtransplantation） (Experimental): The microtransplantation conditioning regimen included high-dose Ara-C chemotherapy (2.0 to 2.5 g/m2 per 12 hours intravenously on days -4 to -2) followed by an infusion of HLA mismatched stem cell 24 hours (day 0) after the completion of cytarabine.
  Interventions: Genetic: HLA mismatched stem cell; Drug: Ara-C
- NST（nonmyeloablative transplantation） (Active Comparator): The NST（nonmyeloablative transplantation）conditioning regimen consisted of 30 mg/m2/d fludarabine for days -6 to -2, 1.5-2 mg/kg/d anti-lymphocyte globulin for days -5 to -2, 40 mg/kg/d cyclophosphamide for days -4 and -2 and 2.0-3.0 g/m2/d cytarabine for days -6 to -4，followed by an infusion of HLA matched stem cell after the completion of regimen. The GVHD prophylaxis included cyclosporine A and mycophenolate mofetil
  Interventions: Genetic: HLA matched stem cell; Drug: cyclosporine A; Drug: Mycophenolate mofetil; Drug: Ara-C; Drug: fludarabine; Drug: anti-lymphocyte globulin; Drug: cyclophosphamide

INTERVENTIONS:
Genetic: HLA mismatched stem cell — HLA mismatched donor G-CSF mobilized peripheral stem cell infused 24 hours (day 0) after the completion of chemotherapy
  Other Names: microtransplantation
  Arms: MST（microtransplantation）
Genetic: HLA matched stem cell — HLA matched donor G-CSF mobilized peripheral stem cell infused after the conditioning reginmen
  Other Names: nonmyeloablative transplantation
  Arms: NST（nonmyeloablative transplantation）
Drug: cyclosporine A — The GVHD prophylaxis included cyclosporine A and mycophenolate mofetil
  Other Names: GVHD prophylaxis
  Arms: NST（nonmyeloablative transplantation）
Drug: Mycophenolate mofetil — The GVHD prophylaxis included cyclosporine A and mycophenolate mofetil
  Other Names: GVHD prophylaxis
  Arms: NST（nonmyeloablative transplantation）
Drug: Ara-C — 2.0 to 3.0g/m2 per 12 hours intravenously for 6 dose
  Other Names: conditioning reginmen
Drug: fludarabine — 30 mg/m2/d for 5days
  Other Names: NST conditioning reginmen
  Arms: NST（nonmyeloablative transplantation）
Drug: anti-lymphocyte globulin — 1.5-2 mg/kg/d for 4 days
  Other Names: NST conditioning reginmen
  Arms: NST（nonmyeloablative transplantation）
Drug: cyclophosphamide — 40 mg/kg/d for 2 days
  Other Names: NST conditioning reginmen
  Arms: NST（nonmyeloablative transplantation）

SUMMARY:
Patients with de novo AML enrolled in the study. Patient who has a HLA-identical donor is assigned to receive NST therapy with GVHD prophylaxis and who has no HLA-identical donor is assigned to receive MST therapy without GVHD prophylaxis.

DETAILED DESCRIPTION:
The optimal therapy for intermediate-risk patients with acute myeloid leukemia (AML) in first complete remission (CR1) is uncertain. Recent studies shown that microtransplantation (MST) can improve survival in AML-CR1 patients. However, a comparison study between the MST and nonmyeloablative stem cell transplantation (NST) is lacking. 156 intermediate-risk AML-CR1 patients aged 9 to 59 years were enrolled in this study. Patients with de novo AML enrolled in the study. Patient who has a HLA-identical donor is assigned to receive NST therapy with GVHD prophylaxis and who has no HLA-identical donor is assigned to receive MST therapy without GVHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have elderly (9-59 ages) AML pathologically confirmed per WHO guidelines.
* Patients WITH intermediate-risk AML-CR1
* Patients must have ECOG Performance status of 0,1,or 2. If ECOG 2.
* Patients must have a HLA mismatched donor who should be able to provide informed consent.
* All genders and races are eligible.
* ALT and AST≤3 ×ULN, TBIL≤1.5 × ULN, Cr≤2 ×ULN or CrCl≥40 mL/min
* By means of ultrasonic Heartbeat map or multiple gated acquisition (MUGA) scanning determination of LVEF in the normal range.
* Donors must be able to safely undergo leukapheresis.

Exclusion Criteria:

* received operation 4 weeks before randomization
* acute promyelocytic leukemia,Myeloid sarcoma, chronic myeloid leukemia in accelerated phase and blastic phase;
* active CNS disease, pregnancy, or other major medical or psychiatric illnesses that could compromise tolerance to this protocol
* Require the use of warfarin or equivalent of vitamin K antagonists (such as phenprocoumon) anticoagulant.
* There is clinical significance of cardiovascular disease, such as uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within 6 months before randomization, or any heart function grade 3 (moderate) or 4 (severe ) heart disease in accordance with the functional classification method of New York Heart Association (NYHA).
* Known to have the following history: human immunodeficiency virus (HIV) or active hepatitis C virus or hepatitis B virus infection
* Any situation processed by the PI that will be damaged to the patients safety.
* Patients and / or authorized family member refuse to sign the consent. attend other clinical researchers in 3 months.
* Donors exclusion criteria include:active infection or malignancy, cardiovascular instability, severe anemia, severe coagulation disorder, pregnancy, inadequate venous access, inability to provide consent, or any other condition deemed unsafe by the treatment staff.

Ages: 9 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2004-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 10 years

SECONDARY OUTCOMES:
treatment-related mortality | 2 years
donor chimerism or microchimerism | 10 years
WT1+CD8+CTL | 10 years
  donor versus leukemia effect
GVHD | 10 years
disease free survival | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: ai huisheng, Principal Investigator — Affiliated Hospital of Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital of Academy of Military Medical Sciences ,, Beijing, Beijing Municipality, China